CLINICAL TRIAL: NCT01957345
Title: Multicentre Evaluation of a New Laboratory Approach for the Diagnosis of Constitutional Functional Disorders of Platelets
Brief Title: Evaluation of a New Approach of the Diagnosis of Constitutional Functional Disorders of Platelets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12 068 08; PHRCI 2012 (Other Grant/Funding Number: French Ministry of Health)
Record Dates: First submitted 2013-06-18; First posted 2013-10-08 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2019-04

CONDITIONS: Platelet Dysfunction
Keywords: constitutional functional disorders of platelets; platelet signalling defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- bleeding disorder (Other): Blood punction at patients with bleeding disorder definitely other than of platelet origin (e.g. "low" von Willebrand)
  Interventions: Other: Blood punction
- constitutional platelet disorder (Other): Blood punction at patients with constitutional platelet disorder (e.g. Glanzmann thrombasthenia)
  Interventions: Other: Blood punction
- defect of platelet function (Other): Blood punction at patients with defect of platelet function of unknown origin, potentially defective in signalling pathway.
  Interventions: Other: Blood punction

INTERVENTIONS:
Other: Blood punction — T1 and T2: one blood punction with signalisation test (T1 for each arm, T2 at +6 months only if an anomaly at signalisation test is detected)
  signalisation test is made by flow cytometry
  Stage 1: for arm "bleeding disorder" : flow cytometry analysis to establish reference values observed in subjects without thrombopathy for each marker after agonist stimulation and corresponding search of an effect if a center-center effect is observed on the reference values its origin will be sought and corrected.
  Stage 2: for the two others arms: Several markers will be analyzed, corresponding to routes or levels of different signaling. For each of these markers, the test will evaluate quantitatively the phosphorylation activity of the protein tested.

SUMMARY:
The primary purpose of the study is to evaluate a standardized method of screening for platelet signalling defects in patients with constitutional disorders of platelet function of unknown origin. We hypothesize that such defects are under-diagnosed in patients, due to heavy workup and requirement of relatively large blood sample by conventional biochemical methods. We propose to analyse kinase signalling downstream platelet membrane receptors using multiplex flow cytometry quantification and fluorescent platelet barcoding.

DETAILED DESCRIPTION:
Little is known of the molecular basis of disorders of signalling pathways potentially responsible of constitutional defects of platelet functions (adhesion, aggregation or secretion) (1-5). Indeed, in routine practice, this investigation is limited by the complexity of the analyse using biochemical methods (western blotting), and the requirement of large amount of platelets.

We have designed a new approach for the quantification of platelet cytoplasmic phosphoproteins by flow cytometry. Fresh platelets in platelet rich plasma are analysed at baseline or after stimulation by major agonists (ADP, TRAP, thromboxane analogue, or collagen-related peptide), with and without relevant inhibitors of each pathway. Multiplex barcoding is used to identify each condition, allowing a high throughput analysis (6, 7). Platelet signalling profiling of Akt, Slp76, P38 MAPK and LIMK can be obtained from a blood sample of less than 10 ml, and within 6h The main objective of the study is to standardize the method between clinical laboratories with a standard expertise in flow cytometry. The study will be performed in 4 academic hospitals members of the French reference network of rare platelet diseases. Three groups of patients referred for mild or severe bleeding disorders will be included: 1) a control group of patients (30 per centre) with a bleeding disorder definitely other than of platelet origin (e.g. "low" von Willebrand); 2) a group of 10 patients per centre with definite constitutional platelet disorder (e.g. Glanzmann thrombasthenia) and 3) a group of 10 patients per centre with a defect of platelet function of unknown origin, potentially defective in signalling pathway.

The control group will serve to standardize the method between centres and to establish the reference values. A quality control will be set up by using frozen platelet preparations. The patients with definite platelet disorder will be useful for detecting potential signalling defects still not described in these pathologies. Platelet signalling defects which could be evidenced in these groups will be further identified by conventional biochemical and molecular methods after confirmation on a new sample.

If this new approach can be proposed to clinical laboratories working on rare platelet diseases, we expect an advance in our knowledge in the field. In addition the method has a potential in pharmaceutical innovation, for identifying (8) or monitoring new antiplatelet agents (9, 10), or identifying platelet defects induced by new "target therapies" designed for other diseases such as cancer or immune pathologies (10).

ELIGIBILITY:
Inclusion Criteria:

* patient consulting for hemorrhagic symptomatology with a bleeding disorder definitely other than of platelet origin (e.g. "low" von Willebrand) / or constitutional platelet disorder (e.g. Glanzmann thrombasthenia) / or with a defect of platelet function of unknown origin, potentially defective in signalling pathway.
* Informed consent form
* patient with social security insurance or equivalent

Exclusion Criteria:

* treatment interfering with platelets function within 7 days prior to enrollment
* thrombocytopenia <100G/L
* pregnant or lactating females
* subjects under juridical protection guardianship or tutelage measure
* subjects involved in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2013-02; Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
standardise the method between clinical laboratories | 3 years
  This is a pilot study of a new approach of screening platelet signalling pathways disorders by flow cytometry with methodological primary outcomes (12) as follows: 1)to standardise the method between clinical laboratories, 2)to establish reference values of the method and 3)to design a quality control assessment
  The primary endpoint will focus on the overall variability of reference values observed in subjects without thrombopathy for each marker after agonist stimulation and corresponding search of an effect if a center-center effect is observed on the reference values its origin will be sought (deviation from the protocol, reagent lot .....) and corrected. The "center effect" will also be analyzed by the quarterly quality control, which will compare the results obtained from the same wafer tests analyzed simultaneously in three sites.

SECONDARY OUTCOMES:
To describe the signalling pathways in platelet disorders | 3 years
  To describe the signalling pathways in platelet disorders with definite diagnosis To screen putative defects in bleeding patients with disorders of platelet function of unknown origin To identify more deeply the defects found in these groups.
  Several markers will be analyzed, corresponding to routes or levels of different signaling. For each of these markers, the test will evaluate quantitatively the phosphorylation activity of the protein tested. We can thus determine for each subject and each marker, the response to the test defined by:
  * The percentage increase in the signal (relative to the rest) after stimulation with a receptor agonist,
  * The percentage increase in the signal (relative to the rest) in the presence of the agonist to the associated receptor antagonist.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SIE, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

REFERENCES:
- [Result] Garcia C, Dejean S, Savy N, Bordet JC, Series J, Cadot S, Ribes A, Voisin S, Rugeri L, Payrastre B, Sie P. Multicolor flow cytometry in clinical samples for platelet signaling assessment. Res Pract Thromb Haemost. 2023 May 16;7(4):100180. doi: 10.1016/j.rpth.2023.100180. eCollection 2023 May. PMID 37538502